CLINICAL TRIAL: NCT05831644
Title: A Randomized, Double-blind, Placebo-controlled, 2-way Cross-over Trial Evaluating the Effect of C21 on Endothelial Dysfunction and Safety in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Trial to Evaluate the Effect of C21 on Endothelial Dysfunction in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vicore Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: VP-C21-013; 2023-000168-77 (EudraCT Number)
Record Dates: First submitted 2023-03-13; First posted 2023-04-26 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Type2diabetes; Endothelial Dysfunction
MeSH Terms: interventions — compound 21

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm 1 (Experimental): A single dose of C21 at visit 2 followed by a single dose of placebo at visit 3.
  Interventions: Drug: C21
- Treatment arm 2 (Experimental): A single dose of placebo at visit 2 followed by a single dose C21 at visit 3.
  Interventions: Drug: C21

INTERVENTIONS:
Drug: C21 — C21 is an angiotensin II type 2 receptor agonist (ATRAG)

SUMMARY:
This trial is a single-centre, randomized, double-blind, placebo-controlled, 2-way cross-over phase 1b trial evaluating the pharmacodynamic effect of C21 on endothelial dysfunction and safety in subjects with type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged ≥ 40 years at the time of the screening visit (Visit 1).
* Documented diagnosed with T2DM prior to the screening visit (Visit 1).
* An RHI score ≤ 2 as assessed by EndoPAT at the time of the screening visit (Visit 1).

Exclusion Criteria:

* Known, active hepatitis B, C, or human immunodeficiency virus (HIV) infection (i.e., HIV with a CD4 (cluster of differentiation 4) count <500 cells/mm³).
* Impaired hepatic function or clinically significant liver disease, which in the investigator's opinion makes the subject inappropriate for this trial.
* Severe renal impairment (i.e., estimated glomerular filtration rate (eGFR) ≤30 mL/min/1.73 m2).
* Prolonged QTcF (QT interval with Fridericia's correction) (>450 ms), atrial fibrillation, clinically significant arrhythmia or other clinically significant abnormality in the resting ECG (electrocardiogram) at screening (Visit 1), as judged by the investigator.
* Unstable or deteriorating cardiac condition.
* Malignancy within the past 5 years with the exception of in situ removal of basal cell carcinoma and cervical intraepithelial neoplasia grade I.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Skånes universitetssjukhus, Malmo, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: C21 First, Then Placebo: Participants first received a single oral dose of C21. After a washout period of 3 to 14 days, they then received a single oral dose of placebo (matching the C21 tablet).
- Experimental: Placebo First, Then C21: Participants first received a single oral dose of placebo (matching the C21 tablet). After a washout period of 3 to 14 days, they then received a single oral dose of C21.
Period: First Intervention
Arm/Group | Experimental: C21 First, Then Placebo | Experimental: Placebo First, Then C21
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Washout Between 1st and 2nd Intervention
Arm/Group | Experimental: C21 First, Then Placebo | Experimental: Placebo First, Then C21
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Experimental: C21 First, Then Placebo | Experimental: Placebo First, Then C21
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: C21 First, Then Placebo | Experimental: Placebo First, Then C21 | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (7.5) | 64.4 (8.5) | 64.5 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pharmacodynamic Effect
Description: Reactive hyperemia index (RHI) score as measured by EndoPAT (Endothelial pulse amplitude tonometry (PAT)). The EndoPAT software, provided with the device, is calculating the RHI using a computerised, automated algorithm.
  Reactive Hyperemia Index (RHI) score is a post-to-pre occlusion pulse amplitude tonometry signal ratio in the occluded arm relative to the same ratio in the control arm, and corrected for baseline vascular tone. RHI is a measure of endothelial function.
  Normal value: RHI > 1.67. Abnormal value: RHI ≤ 1.67. There is no theoretical minimum and/or maximum values for the RHI score.
  A lower RHI score following C21 compared to placebo is the desired outcome.
Time Frame: Maximum 15 days after first Investigational Medical Product (IMP) intake.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- C21 Treatment: Subjects received a single dose of 200 mg C21 (4 oral capsules) at Visit 2 or Visit 3.
- Placebo Treatment: Subjects received a single dose (4 oral capsules) of placebo at Visit 2 or Visit 3.
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 11 | 11
score on a scale | 1.787 (0.062) | 1.911 (0.062)
Statistical Analysis 1: Comparison: C21 Treatment vs Placebo Treatment; The primary endpoint (RHI score) was compared between treatments using an analysis of variance model (ANOVA) with treatment and period as fixed effects and subjects as random effect; Test type: Superiority; p = 0.1925, ANOVA; Mean Difference (Final Values) = -0.124, 90% CI 2-sided [-0.285 to 0.037]

2. Secondary Outcome: Augmentation Index (AI) Score as Measured by EndoPAT (Endothelial Pulse Amplitude Tonometry (PAT)). The AI Score Reported is Change Between Baseline Value and Value at the Visit Where Either C21 or Placebo is Taken.
Description: The EndoPAT software, provided with the device is calculating the the Augmentation index (AI) using a computerised, automated algorithm. Augmentation index is a measurement of vascular stiffness. Augmentation index is calculated from PAT pulses based on the following formula AIx = 100 × (Augmentation pressure)/(Pulse Pressure). Ideally the augmentation index is somewhere between 20-80, but can be both negative and positive depending on the value of the augmentation pressure. A higher value is indicative of vascular stiffness.
Time Frame: Maximum 15 days after first Investigational Medical Product (IMP) intake.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 11 | 11
score on a scale | 15.937 (2.484) | 20.877 (2.484)
Statistical Analysis 1: Comparison: C21 Treatment vs Placebo Treatment; The secondary pharmacodynamic endpoint (AI) was analysed using a similar ANOVA model as for the primary endpoint; Test type: Superiority; p = 0.1941, ANOVA; Mean Difference (Final Values) = -4.940, 90% CI 2-sided [-11.392 to 1.513]

ADVERSE EVENTS:
Time Frame: All events meeting the definition of an AE was reported in the period from the subject has signed the informed consent form (screening visit) until the end-of-trial visit. Depending on visit schedule this period can be up to 49 days.
Arm/Group | C21 Treatment | Placebo Treatment
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 2/11 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C21 Treatment (N=11) | Placebo Treatment (N=11)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT05831644/Prot_SAP_000.pdf